CLINICAL TRIAL: NCT02226900
Title: Myocardial Hybrid Revascularization Versus Coronary artERy Bypass GraftING for Complex Triple-vessel Disease
Acronym: MERGING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: InCor Heart Institute (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Pedro A. Lemos, Pedro A. Lemos, Professor of Medicine, InCor Heart Institute, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MERGING
Record Dates: First submitted 2014-08-21; First posted 2014-08-27 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Multivessel Coronary Artery Disease
Keywords: Multivessel Coronary Artery Disease; Hybrid Revascularization
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hybrid Revascularization (Experimental): The hybrid myocardial revascularization group will be accomplished by a two-step scheme, comprised by off-pump LIMA-to-left anterior descending grafting, followed by percutaneous coronary interventions with Promus Element (everolimus second generation drug eluting stent) for the remaining coronary lesions.
  Interventions: Procedure: Hybrid Revascularization
- Conventional Surgical Coronary Bypass Grafting (Other): Conventional Coronary Artery Bypass Grafts with in pump technique.
  Interventions: Procedure: Conventional Coronary Artery Bypass Surgery

INTERVENTIONS:
Procedure: Hybrid Revascularization — Off-pump LIMA connected to the left anterior descending artery followed by percutaneous coronary intervention with drug eluting stents to the other territories.
  Arms: Hybrid Revascularization
Procedure: Conventional Coronary Artery Bypass Surgery — On pump coronary artery by-pass surgery
  Other Names: Surgery
  Arms: Conventional Surgical Coronary Bypass Grafting

SUMMARY:
This is a pilot randomized study that aim to assess the safety and feasibility of a hybrid myocardial revascularization strategy (coronary artery by-pass graft and percutaneous intervention) in comparison with conventional surgical coronary bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

* Triple-vessel disease with proximal or mid LAD disease with angiographic diameter stenosis > 70% by visual analysis in all three territories, requiring myocardial revascularization OR triple-vessel disease with proximal or mid LAD disease with angiographic diameter stenosis 50-70% by visual analysis in any territory but with invasive or non-invasive evidence of flow-limiting stenosis in all three territories, requiring myocardial revascularization
* Total SYNTAX score > 22
* LCx and RCA territories estimated to be equivalently revascularized by either PCI or CABG, with at least one major non-LAD vessel to be treated
* Clinical and anatomic eligibility for both PCI and CABG as agreed to by both interventional and surgical consensus

  * Interventionalist determines PCI appropriateness and eligibility
  * Surgeon determines surgical appropriateness and eligibility
* Silent ischemia, stable angina, unstable angina or recent MI

  * If recent MI, cardiac biomarkers must have returned to normal prior to randomization
* Ability to sign informed consent and comply with all study procedures

Exclusion Criteria:

* Prior PCI or CABG at any time prior to randomization
* Need for any concomitant cardiac surgery other than CABG (e.g. valve surgery, aortic repair, etc.), or intent that if the patient randomizes to surgery, any cardiac surgical procedure other than isolated CABG will be performed
* Patients unable to tolerate, obtain or comply with dual antiplatelet therapy for at least one year
* Patients requiring additional surgery (cardiac or non cardiac) within one year
* The presence of any clinical or anatomical condition(s) which leads the participating interventional cardiologist to believe that clinical equipoise is not present (i.e. the patient should not be treated by PCI, but rather should be managed with CABG or medical therapy - reasons will be documented)
* The presence of any clinical or anatomical condition(s) which leads the participating cardiac surgeon to believe that clinical equipoise is not present (i.e. the patient should not be treated by CABG, but rather should be managed with PCI. or medical therapy - reasons will be documented)
* Non cardiac co-morbidities with life expectancy less than 1 year
* Other investigational drug or device studies that have not reached their primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Revascularization Procedure Proposed by the Heart Team | 30 days
  The primary endpoint of this pilot study is the feasibility of revascularization planned preoperatively by the Heart team in the absence of adverse events (death, myocardial infarction, stroke, or unplanned revascularization) at 30 days.

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events | 1 year
  Composite and isolated measure of adverse events (all-cause death, myocardial infarction, stroke, or unplanned revascularization) at 1 year and annually up to 5 years.
Major Adverse Cardiovascular Events | 2 years
  Composite and isolated measure of adverse events (all-cause death, myocardial infarction, stroke, or unplanned revascularization) at 1 year and annually up to 5 years.
Major Adverse Cardiovascular Events | 3 years
  Composite and isolated measure of adverse events (all-cause death, myocardial infarction, stroke, or unplanned revascularization) at 1 year and annually up to 5 years.
Major Adverse Cardiovascular Events | 4 years
  Composite and isolated measure of adverse events (all-cause death, myocardial infarction, stroke, or unplanned revascularization) at 1 year and annually up to 5 years.
Major Adverse Cardiovascular Events | 5 years
  Composite and isolated measure of adverse events (all-cause death, myocardial infarction, stroke, or unplanned revascularization) at 1 year and annually up to 5 years.
Major Adverse Cardiovascular Events | 180 days
  Composite and isolated measure of adverse events (all-cause death, myocardial infarction, stroke, or unplanned revascularization) at 1 year and annually up to 5 years.
Safety | 1 year
  Cause of death (cardiac vs. non-cardiac); MI type; stroke type and severity.
Recurrence of Angina | 1 year
  Analyse patient recurrence of angina according to the Canadian Cardiovascular Society (CCS)
Medication Impact | 1 year
  Impact of antithrombotic agents and dual antiplatelet therapy in peri-procedural and long-term follow up safety end points.
Stent Thrombosis | 1 year
  Evaluate stent thrombosis according to the ARC (Academic Research Consortium) criteria
Bleeding | 1 year
  Hemorrhagic complications according to the BARC (Bleeding Academic Research Consortium) criteria
Neurological Events | 1 year
  Evaluate neurological complications by clinical tests (physical examination), vascular ultrasound and doppler perfusion measures.
Graft Patency | 1 year
  Patency of grafts and coronary artery disease at 1 year of follow-up evaluated by angiotomography
Clinical and Angiographic Scores Correlation with Prognostic | 1 year
  Evaluate the clinical correlation between the revascularization strategy and the usefulness of the SYNTAX score, ACEF score, clinical SYNTAX score, logistic EuroSCORE, STS score and InsCor for prognostic evaluation
Efficacy of the Strategy | 1 year
  Evaluate and compare the rate of repeated revascularization (target lesions and target vessels) in each one of both strategies.
Symptomatic Graft Occlusion | 1 Year
  Evaluate patients that presented with recurrent ischaemia symptoms due to graft occlusion. The diagnostic must be done by angiography or angiotomography.

OTHER OUTCOMES:
Quality of life. | 5 years
Cost | 5 years
  Evaluate and compare the final cost of the procedure and follow up period of the patients enrolled in each one of the strategies.
Hospital Stay | 1 year
  Evaluate and compare the period of hospital stay of the patients enrolled in each one of the strategies.

CONTACTS AND LOCATIONS:
Locations (1):
- InCor -Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil